CLINICAL TRIAL: NCT00989313
Title: A 12 Month, Long-term Follow-up Study of Patients With Actinic Keratosis on Non-head Locations (Trunk and Extremities) Who Have Completed Day 57 in Study PEP005-028 (REGION Ib)
Brief Title: A Long Term Follow up Study of Patients Who Have Complete Clearance of Their Actinic Keratosis (AK) Lesions at the Day 57 Visit in the PEP005-028 Study
Status: Completed | Type: Observational
Sponsor: Peplin (Industry)
Responsible Party: Sponsor
Other Study IDs: PEP005-032
Record Dates: First submitted 2009-10-01; First posted 2009-10-05 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Actinic Keratosis
Keywords: Peplin; Actinic keratosis; PEP005
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Drug: Lesion count

INTERVENTIONS:
Drug: Lesion count — Lesion count in area treated by study drug in a prior study. No drug will be applied during this long-term follow up study. Drug was applied during the primary study.
  Other Names: AK lesion recurrence

SUMMARY:
This study is designed to follow up patients, who have participated in the PEP005-028 study and observed complete clearance of their Actinic Keratosis (AK) lesions, over a 12 month period to assess both recurrence of AK lesions and long term safety in the selected treatment area.

ELIGIBILITY:
Inclusion

* Patient has provided informed consent documented by signing the Informed Consent Form (ICF) prior to any study-related procedures
* Patient achieved complete clearance of AK lesions (lesion count of 0) in the selected treatment area at the Day 57 visit in the following Peplin AK clinical Study: PEP005-028

Exclusion

* Concurrent participation in another research study which would involve the selected treatment area (except for any post-study follow-up visits for previous Peplin AK study)
* Early termination from study PEP005-028

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who achieved complete clearance of AK lesions at the Day 57 visit in the PEP005-028 study
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2009-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Summarize treatment area recurrence of AK lesions, in the selected treatment area during a 12 month follow-up period for patients with complete clearance, who have completed Day 57 in Study PEP005-028. | 12 months

SECONDARY OUTCOMES:
Summarize long-term safety data, in the selected treatment area over a 12 month follow-up period for patients with complete clearance, who have completed Day 57 in Study PEP005-028. | 12 months

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Burke Pharmaceutical Research, Hot Springs, Arizona
  - Skin Surgery Medical Group Inc., San Diego, California
  - Atlanta Dermatology, Vein & Research Center, LLC, Alpharetta, Georgia
  - Altman Dermatology Associates, Arlington Heights, Illinois
  - Glazer Dermatology, Buffalo Grove, Illinois
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Skin Specialists, PC, Omaha, Nebraska
  - Karl G. Heine Dermatology, Henderson, Nevada
  - Group Health Associates, Cincinnati, Ohio
  - DermResearch, Inc., Austin, Texas
  - Suzanne Bruce and Associates, PA, The Center for Skin Research, Houston, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Dermatology Associates of Tyler, Tyler, Texas
  - Dermatology Research Centre, Salt Lake City, Utah
  - The Education and Research Foundation, Lynchburg, Virginia
  - Virginia Clinical Research, Inc, Norfolk, Virginia

REFERENCES:
- [Derived] Lebwohl M, Shumack S, Stein Gold L, Melgaard A, Larsson T, Tyring SK. Long-term follow-up study of ingenol mebutate gel for the treatment of actinic keratoses. JAMA Dermatol. 2013 Jun;149(6):666-70. doi: 10.1001/jamadermatol.2013.2766. PMID 23553119
- See also: Food and Drug Authority — http://www.fda.gov